CLINICAL TRIAL: NCT05016869
Title: A Phase Ⅰb/Ⅱ Study of Fruquintinib Combined With Capecitabine in the First-line Maintenance Treatment of RAS/BRAF Wild-type Metastatic Colorectal Cancer
Brief Title: Fruquintinib Plus Capecitabine as Maintenance Treatment of RAS / BRAF Wild-type Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Lin Yang, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C102
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): fruquintinib plus capecitabine
  Interventions: Drug: fruquintinib plus capecitabine

INTERVENTIONS:
Drug: fruquintinib plus capecitabine — Ⅰb: capecitabine: 1000 mg/m²，PO BID, d1-14，Q3W; fruquintinib 3mg/4mg/5mg, d1-14, PO QD, Q3W.
  ⅠⅠ: fruquintinib RP2D, d1-14, PO QD, Q3W, capecitabine: 1000 mg/m²，PO BID, d1-14，Q3W

SUMMARY:
This phase I/II study was designed to evaluate the efficacy and safety of fruquintinib combination with capecitabine in maintenance treatment after first-line chemotherapy combined with cetuximab.

DETAILED DESCRIPTION:
At present, most studies use chemotherapy combined with cetuximab or cetuximab alone as the maintenance treatment scheme after the first-line regimen containing cetuximab. However, the skin reaction caused by cetuximab and frequent infusion treatment will bring inconvenience to patients. MACBETH study compared the maintenance of bevacizumab with cetuximab, although there was no significant difference in PFS between them, the Bev group seemed to convey a longer median OS. Fruquintinib is a highly selective anti angiogenesis TKI. This study aims to explore the efficacy and safety of fruquintinib combined with capecitabine in maintenance treatment after first-line chemotherapy combined with cetuximab. Both fruquintinib and capecitabine are orally given, so this regimen may provide a maintenance treatment option that is more manageable for patients in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic colorectal adenocarcinoma;
* 18-75 years old;
* Eastern Cooperation Oncology Group (ECOG) performance score 0-1;
* At least one evaluable lesion for disease assessment according to RECIST version 1.1;
* Able to take oral medications;
* Patient have achieved CR, PR or SD after up to 8 cycles of first-line standard FOLFOX / - FOLFIRI / XELOX / xeliri + cetuximab treatment, and remained unresectable;
* If radiotherapy has been performed before enrollment, at least one lesion should be located outside the radiation field;
* Adequate organ functions as assessed by the following laboratory requirements: Leukocytes≥3.0x10^9/L, absolute neutrophil count≥1.5x10^9/L, platelet count≥100x10^9/L, hemoglobin≥9g/dL; serum bilirubin≤1.5x the upper limit of normal(ULN);Alanine aminotransferase(ALT) and aspartate aminotransferase(AST)≤2.5x ULN; serum creatinine≤1.5x ULN.
* An expected survival of at least 12 weeks;
* Fertile male or female patients volunteered to use effective contraceptive methods during the study period and within 6 months after the end of treatment;
* Willing to provide written informed consent to study procedures.

Exclusion Criteria:

* Patients who have received fruquintinib;
* Patients who have received TACE within 6 weeks before enrollment;
* Participated in other unapproved or unlisted drug clinical trials in China within 4 weeks before enrollment, and received corresponding experimental drug treatment;
* Patients with dysphagia, active peptic ulcer, intestinal obstruction, active gastrointestinal bleeding, peptic perforation, malabsorption syndrome or uncontrolled intestinal inflammatory diseases;
* International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 × ULN；
* The researchers judged clinically significant electrolyte abnormalities;
* At present, the patient has hypertension that cannot be controlled by drugs, which is specified as: systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg;
* Patients currently have poorly controlled diabetes (fasting glucose level is greater than CTCAE grade 2 after regular treatment);
* Have received any surgery or invasive treatment or operation within 4 weeks before enrollment (except venous catheterization, puncture and drainage, etc.);
* Active or uncontrolled severe infection ≥ grade 2 according to National Cancer Institute Common Toxicity (NCI-CTC) criteria;
* Uncontrolled central nervous system metastasis or previous brain metastasis;
* Other malignant tumors in the past 5 years, except for skin basal cell or squamous cell carcinoma after radical surgery, or cervical carcinoma in situ;
* Any kind of concurrent cardiac disease with clinical meanings, such as cardiovascular accident, myocardial infarction, thromboembolism or hemorrhage within 6 months before enrollment, congestive heart failure ≤New York Heart Association (NYHA) class 2; ventricular arrhythmias requiring drug treatment; LVEF < 50%;
* With positive urine protein and 24-hour urinary protein content>1g;
* Have a tendency of bleeding or clotting;
* Known human immunodeficiency virus (HIV) infection; known history of clinically significant liver disease, including viral hepatitis;
* The target lesions have received brachytherapy (radioactive particle implantation) within 60 days before admission;
* Unrelieved toxic reactions higher than CTCAE V5.0 grade 1 caused by any previous anti-cancer treatment, excluding hair loss, lymphopenia and neurotoxicity ≤ grade 2 caused by oxaliplatin;
* With any illness or medical conditions that may jeopardize the patient's compliance or interfere the analyses or judgements of study results;
* Pregnancy or lactation at the time of study entry;
* With fertility but refuse to contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
recommended phase 2 dose (RP2D) | up to 1 year
  RP2D is determined according to DLT and MTD in the phase 1 study
progression-free survival (PFS) | up to 3 years
  PFS is defined as the time from the start of maintenance treatment to the earliest evidence of disease progression (per RECIST v1.1), or death from any cause

SECONDARY OUTCOMES:
disease control rate (DCR) | up to 3 years
  DCR is defined as the proportion of patients achieving complete response, partial response or having stable disease
objective response rate (ORR) | up to 3 years
  ORR is defined as the proportion of patients achieving complete response or partial response
overall survival (OS) | up to 3 years
  OS is defined as the time from randomized to death from any cause or to last contact
Adverse events (AEs) | up to 3 years
  Adverse events assessments are computed and categorized according to the Common Toxicity Criteria of the National Cancer Institute, version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- National Center/Cancer Hospital, China Academy of Medical Science and Peking Union Medical College, Beijing, China